CLINICAL TRIAL: NCT01906398
Title: Evaluation of the Efficacy and Safety of Ketogenic Diet as Adjunctive Treatment in Adults With Refractory Epilepsy: a Pilot Study.
Brief Title: Efficacy and Safety of Ketogenic Diet as Adjunctive Treatment in Adults With Refractory Epilepsy
Acronym: KD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mid-Atlantic Epilepsy and Sleep Center, LLC (Other)
Responsible Party: Principal Investigator, Pavel Klein, MD, Mid-Atlantic Epilepsy and Sleep Center, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: maes 001
Record Dates: First submitted 2013-06-11; First posted 2013-07-24 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Epilepsy
Keywords: Refractory epilepsy; ketogenic diet; efficacy
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: ketogenic diet (Other): Treatment will consist of KD will consist of 3:1 [fat]: [protein + carbohydrate] weight ratio, with 1600 kcal restriction for patients with body mass index (BMI) of ≥ 21. The diet will be initiated with a 24 hour fast to induce ketosis. The diet will be supplemented with vitamins, calcium and phosphorus supplements to meet the requirements of US Dietary Reference Intakes (DRI) standard. If seizure frequency does not improve after 3 months of KD treatment, [fat]: [protein + carbohydrate] weight ratio will be increased to 4:1
  Interventions: Other: ketogenic diet

INTERVENTIONS:
Other: ketogenic diet — KD will consist of 3:1 [fat]: [protein + carbohydrate] weight ratio, with 1600 kcal restriction

SUMMARY:
The purpose of the study is to obtain pilot data on safety and efficacy of ketogenic diet (KD) as adjunctive treatment of adults with refractory epilepsy. This will be an open label study comparing seizure frequency during 4 months of prospective baseline observation period with seizure frequency during 4 months of add-on KD treatment. 18-65 year old men and women with refractory epilepsy, defined as seizures persisting in spite of past/present treatments with ≥ 3 AEDs, with seizure frequency of ≥ 0.5/month, will be evaluated. Subjects with both primary generalized and localization-related epilepsy (PGE, LRE) will be recruited. Subjects will have had epilepsy for at least 2 years prior to enrollment. Following initial screening, subjects will be observed for 4 months, with no change in AEDs except when deemed necessary by the patient's neurologist according to standard clinical care. Patients will then start ketogenic diet. Evaluations will include seizure frequency using a seizure diary, adverse events, treatment compliance using urine and plasma ketone levels. Quality of life will be evaluated with a standardized questionnaire of Quality Of Life In patients with Epilepsy, QOLIE-31-P. Level of alertness will be evaluated with Epworth Sleepiness Scale. These questionnaires will be administered at each visit.

DETAILED DESCRIPTION:
The goal of the present open label study is to obtain pilot data to evaluate the efficacy and safety of KD in adults with intractable epilepsy. Investigators will evaluate the effect of KD on seizure frequency and on adverse events. Investigators will also evaluate serum levels of the ketone body, βhydroxybutyrate (BOH) and of glucose in order to determine whether changes in serum levels of these substances correlate with KD-associated changes in seizure frequency. The data from the present study will be used to design a large randomized study.

Laboratory evaluations will include complete blood count (CBC), serum electrolytes, including calcium, phosphate and magnesium, renal and liver functions, including total protein and albumin, uric acid, fasting serum lipid profile, glucose and b- hydroxybutyrate (BOH) levels, serum carnitine level, serum a.m. trough antiepilepsy drugs levels, and urine calcium and creatinine level. They will be obtained twice at baseline a month apart and monthly during KD treatment.

Primary outcome measures will include average monthly seizure frequency and adverse events. Secondary outcome measures will include treatment compliance, quality of life questionnaire (QOLIE-31-P) scores, and Epworth Sleepiness Scale scores.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Stable epilepsy, either primary generalized or localization-related with partial complex seizures including partial complex seizures with or without secondary generalization, partial simple seizures with a clear motor component with or without secondary generalization, and partial simple seizures with secondary generalization; primary generalized tonic clonic seizures; and absence seizures of > 10 sec duration.
3. Stable AED doses for at least 30 days
4. Epilepsy duration for > 1 year
5. Past/current treatment with > 3 AEDs. Vagal nerve stimulation treatment will be allowed and will not count as an AED. Vagal nerve stimulation setting must be stable for 3 months prior to enrollment
6. Seizure frequency of > 0.5/month

Exclusion Criteria:

1. Exclusively myoclonic seizures or absence seizures of ≤ 10 sec duration; simple partial seizures without motor components or secondary generalization
2. Non-epileptic seizures
3. Progressive neurological disease including neoplasm, central nerve system degenerative disorders including Alzheimer's disease, other forms of dementia
4. Any systemic illness or unstable medical condition that might pose additional risk, including: renal or liver disease, past history of renal calculi, hyperuricemia, hypercalcemia, mitochondrial disease, known disorder of fatty acid metabolism, porphyria, other unstable metabolic or endocrine disturbances, and active systemic cancer
5. Familial hyperlipidemia or uncontrolled hyperlipidemia
6. Body Mass Index (BMI) < 18
7. Change in the dose of any Antiepileptic Drug within 30 days prior to enrollment
8. Psychosis within six months of enrollment.
9. Active drug or alcohol dependence or any other factors that, in the opinion of the site investigators would interfere with adherence to study requirements;
10. Pregnancy
11. Use of any CNS-active investigational drugs within 3 months of enrollment.
12. Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in epileptic seizure frequency. | baseline, 8 months
  Seizure frequency, adverse events and treatment compliance will be reviewed. The diet will be reviewed with the subject by the nutritionist before treatment initiation. Seizure frequency will be counted using a daily seizure diary. Subject's neurological and other clinical progress since the last visit will be reviewed. Concurrent medications will be documented. Vital signs and weight will be obtained, and a complete physical and neurological examination will be performed. Body mass index will be calculated. Subjects seizure/urine ketone diary will be reviewed at each visit.
  Treatment compliance will be evaluated with urine ketone levels using the diaries and with serum b-hydroxy-butyrate (b-OH-butyrate, BOH) levels.

SECONDARY OUTCOMES:
Evaluate the number of participants with adverse events. | baseline, 8 months
  Adverse events and treatment compliance will be reviewed.Subject's neurological and other clinical progress since the last visit will be reviewed.

OTHER OUTCOMES:
Changes from baseline in Quality of life. | baseline, 8 months
  Quality of life will be evaluated with a standardized questionnaire of quality of life in patients with epilepsy, QOLIE-31-P.
Changes from baseline in alertness. | baseline, 8 months
  Alertness will be evaluated with Epworth Sleepiness Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Klein, MD, Principal Investigator — Mid-Atlantic Epilepsy and Sleep center
Locations (1):
- MidAtlantic Epilepsy and Sleep Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided